CLINICAL TRIAL: NCT01810419
Title: Estimation of Spleen Size With Hand Held Ultrasound
Brief Title: Ultrasound Estimation of Spleen Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Graydon Meneilly, MD, FRCPC, FACP, Professor & Eric W. Hamber Chair, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H12-03055
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Splenomegaly
Keywords: splenomegaly; ultrasound; Vscan
MeSH Terms: conditions — Splenomegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- normal and various degrees splenomegaly (Experimental): Vscan Ultrasound (GE Healthcare, USA) Conventional Ultrasound (Ultrasonix) used to determine spleen size Crossover design, all subjects will be measured with both devices. half will have the handheld done first, then conventional half the Conventional done first, then handheld
  Will complete questionaire for both:
  1. Adequacy of image quality
  2. What is best view obtained
  3. Greatest Longitudinal Measure
  4. Diagnosis
  5. Diagnostic Certainty
  6. Time to Complete exam
  Interventions: Device: Vscan Ultrasound (GE Healthcare, USA); Device: Conventional Ultrasound

INTERVENTIONS:
Device: Vscan Ultrasound (GE Healthcare, USA) — Vscan Ultrasound used to determine spleen size and the other qualities described in the arm description.
  Other Names: handheld ultrasound (HCU)
Device: Conventional Ultrasound — Conventional Ultrasound used to determine spleen size and the other qualities described in the arm description.
  Other Names: Gold standard; standard ultrasound; Ultrasonix

SUMMARY:
In internal medicine, assessment of spleen size on physical examination is an extremely important part of the overall evaluation of patients with many illnesses. Examination of the spleen is also one of the core competencies that the investigators expect our students and residents to learn as part of their training. Unfortunately, the sensitivity and specificity of examination of the spleen at the bedside is not very good. The investigators wish to determine if handheld ultrasound can accurately assess spleen size. Doing so would make physical examination of the spleen obsolete and transform training objectives for medical students and residents.

DETAILED DESCRIPTION:
The diagnosis of splenomegaly (abnormal enlargement of the spleen) is extremely important in managing patients with many medical conditions. The ability to recognize an enlarged spleen in a timely manner can impact patient outcomes. Although the physical exam can be used to confidently diagnosis massive enlargement of the spleen, evaluating lesser degrees of splenomegaly at the bedside proves more difficult. In current practice, the gold standard for diagnosis of splenomegaly is the standard abdominal ultrasound. The prevalence of splenomegaly in patients with several medical conditions such as blood disorders and cirrhosis is relatively high. Therefore, the demand for abdominal ultrasound is evergrowing and similarly the cost of caring for patients with these diseases increases.

Examination of the spleen is one of the core competencies that we expect our students and residents to learn as part of their training. This physical diagnosis manoeuver is frequently used to examine residents at the Royal College level and determine their fitness to practice. Unfortunately, the sensitivity and specificity of examination of the spleen at the bedside is not very good.

With the introduction of handheld ultrasound (HCU) devices, rapid bedside assessment of a patient is now possible. The Pocket-sized Vscan Ultrasound device (Vscan) (GE Healthcare, USA) allows for 2D imaging on a 3.5 inch display and has been shown to have comparable image quality to standard ultrasound for some applications. The Vscan and other HCU devices have been used at point of care to evaluate a number of conditions and can greatly impact treatment decisions in medical patients at the bedside. The ability to recognize splenomegaly in a timely manner can impact patient outcomes. In addition, the use of this technology could significantly impact training standards for students and residents.

It remains unclear whether bedside evaluation with the Vscan is able to accurately measure spleen size. Our study aims to determine the diagnostic accuracy of the Vscan when used by trained ultrasonographers, in patients with varying degrees of splenomegaly. If we can reliably show that a trained ultrasonographer can accurately characterize spleen size at the bedside with a handheld device, the next stage of the study will involve training medical residents in the use of handheld ultrasound to see if they can also reliably assess spleen size.

ELIGIBILITY:
Inclusion Criteria:

* patients in the practices of hematologists at VGH (Vancouver General Hospital) who are expected to have normal size spleens as well as various degrees of splenomegaly

Exclusion Criteria:

* will exclude patients who cannot speak English or who cannot give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
longitudinal measure of spleen in centimeters | 1 day

SECONDARY OUTCOMES:
Diagnosis of spleen size | 1 day
  Diagnosis
  1. No Splenic Enlargement
  2. Moderate Splenic Enlargement
  3. Massive Splenic enlargement
time to complete Vscan examination | 1 day
  Time to complete Vscan exam
  1. <5min
  2. 5-10 min
  3. 10-15min
  4. >15min

OTHER OUTCOMES:
Image quality and best views | 1 day
  Adequacy of study
  1. Image quality inadequate to make diagnosis
  2. Image quality adequate
  3. Image quality excellent
  Best Views obtained
  1. Supine
  2. Right Lateral Decubitus
Diagnostic Certainty | 1 day
  Diagnostic Certainty
  1. Not confident
  2. Somewhat confident
  3. Very confident

CONTACTS AND LOCATIONS:
Overall Officials: Graydon S Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health (VCHRI/VCHA), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No